CLINICAL TRIAL: NCT04110600
Title: Efficacy of Coffee Versus Peppermint Oil Intake in Promoting GIT Motility After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, amaal ehab mostafa, obstetrics and gynaecology resident, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FWA000017585
Record Dates: First submitted 2019-09-21; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Gastrointestinal Motility and Defecation Conditions
Keywords: Bowel movements; Cesarean section; Oral hydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coffee group (Active Comparator): This group includes 300 patients who underwent cesarean delivery under spinal anaesthesia And will have 100 ml of coffee after 2,4 and 6 hours
  Then outcomes will be assessed as per time frame
  Interventions: Other: Coffee effect on early gastric motility
- Pepper mint oil group (Active Comparator): This group includes 300 patients who underwent cesarean delivery under spinal anaesthesia This group will have 100 ml of pepper mint oil After 2,4 and 6 hours
  Then outcomes will be assessed as per time frame
  Interventions: Other: Efficacy pepper mint oil on motility

INTERVENTIONS:
Other: Coffee effect on early gastric motility — this group 100ml coffee after two hours
  Other Names: Coffee intake
  Arms: Coffee group
Other: Efficacy pepper mint oil on motility — This group 100me pepper mint oil after 2 hours
  Other Names: Pepper mint oil
  Arms: Pepper mint oil group

SUMMARY:
It is a comparison between coffee effect versus peppermint oil in promoting GIT motility after cesarean section

DETAILED DESCRIPTION:
This study includes 600 patients who underwent cesarean delivery under spinal anaethesia subdivided into two groups each contain 300 patients Group 1 will have 100 ml of coffee after 2,4 and 6 hours Group 2 will have 100 me of pepper mint oil After 2,4 and 6 hours

Then outcomes will be assessed as per time frame

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate.
* uncomplicated pregnancy.
* uncomplicated cesarean section.
* under regional anesthesia
* BMI<30kg/m.
* level of hemoglobin is 10g/dl or more

Exclusion Criteria:

* medical disorders in the form of HTN,DM and hepatic disorders and bleeding disorders
* intra operative bowel or bladder injury during the cesarean section
* intra operative severe bleeding
* chronic gastrointestinal problems like chronic constipation ,peptic ulcer ,esophagitis ,hiatus hernia and IBS
* sever intestinal adhesions
* Respiratory problems and infection that require medication intervention
* operation more than 90 minutes

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Regain of GIT motility after cesarean section by auscultation of intestinal sound | First 12 hours after cs
  Auscultation of intestinal sounds hourly for first 12. Hours

SECONDARY OUTCOMES:
Sense of nausea | First 24 hours after cs
  Nausea sensation
Sense of vomiting | First 24 hours after cs
  Recording time for first time of vomiting
First passage of flatus | First 24 hours after cs
  Record first passage of flatus
First defection | First 24 hours after cs
  Record first bowel motjon
Effect on abdominal distention | First 24 hours after cs
  Recording incidence of distension
Need of medication to enhance motility of GIT | First 24 hours after cs
  Assessing need for extra medications for motility
Length of hospital stay after surgery | First 24 hours after cs
  Recording length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Nermine Elghareb, Lecturer, Study Director — Ain Shams Maternity Hospital; Ahmed Tharwat, Professor, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No